CLINICAL TRIAL: NCT05515497
Title: BMT4me: Improving Adherence Through mHealth for Pediatric Stem Cell Transplant Patients (BMT4me 2.0)
Brief Title: BMT4me: Post-HSCT Medication Adherence mHealth App
Acronym: Bmt4me 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Micah Skeens (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Micah Skeens, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002478; 4R00NR019115-03 (NIH)
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Stem Cell Transplant; Adherence, Medication; Digital Health
Keywords: Adherence; mHealth; Stem Cell transplant; Immunosuppression; Digital Health; Pediatrics
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BMT4me 2.0 Intervention Group (Experimental): The intervention group will be receiving the BMT4me 2.0 app at discharge as the primary intervention.
  Interventions: Device: BMT4me 2.0 app
- BMT4me 2.0 Control Group (No Intervention): The control group will be receiving usual care at discharge. These participants will not be receiving the BMT4me 2.0 app.

INTERVENTIONS:
Device: BMT4me 2.0 app — The BMT4me app was designed by AWRI RISI developers and has been through multiple phases of stakeholder testing. The app is a virtual assistant for caregivers, allowing for medication record keeping, medication and refill reminders, symptom tracking, and a word and picture journal. All data is secured on the individuals password protected phone.
  Arms: BMT4me 2.0 Intervention Group

SUMMARY:
This is a mixed methods, prospective longitudinal pilot RCT to evaluate the 1) acceptability of a newly developed mHealth app (BMT4me), 2) the feasibility of enrolling and retaining caregivers of children in the acute phase post-HSCT, and 3) the potential efficacy of an mHealth app on adherence to immunosuppressants in post-HSCT children discharged during the acute phase.

DETAILED DESCRIPTION:
In the United States, poor adherence accounts for up to 70% of all medication-related hospital admissions, resulting in $100 billion in healthcare costs annually Adherence rates have been reported as low as 0% in pediatric patients. Reasons for non-adherence are multifactorial. The most important determinants of non-adherence are consistently documented as complexity and duration of treatment regimens, as well as forgetfulness. Thus, children undergoing difficult hematopoietic stem cell transplants (HSCT) that require medication indefinitely are at high risk for medication non-adherence.

Only 4 published studies exist regarding adherence in pediatric HSCT. None address adherence to immunosuppressant medication, nor are they RCTs. Second, the complexity of most interventions for adherence is counter to the geographic, resource, and time constraints families of chronically ill children face. Adherence interventions based on conventional behavior theory have been cumbersome for families already stressed due to chronic illness. BE design is a significant paradigm shift to a simpler, less onerous approach that can engage those patients and families that would otherwise forego complicated adherence interventions. Although mHealth adherence apps are a widely available, simple, and innovative approach to addressing these problems, a third gap relates to poor usability. For example, a recent review of pediatric adherence apps found that none identified individual barriers to adherence, and nearly all were designed for adults. Thus, there is an urgent need to develop and evaluate innovative, accessible, and evidence-based approached to adherence among children receiving HSCT to prevent morbidity and mortality from GVHD.

The impact of non-adherence on clinical outcomes is largely unknown in pediatric HSCT. poor adherence is generally associated with adverse outcomes, including complications, hospital admissions, and even death. The societal burden of cancer care and HSCT is substantial and likely to increase based on the growing number of transplants each year. Clinicians and researchers have focused on GVHD prevention to minimize unnecessary treatment-related deaths. Acute GVHD develops in the first 100 days post-transplant. Children that develop acute GVHD have a 30% to 50% chance of survival. Morbidity and mortality due to GVHD can be decreased through prophylactic use of immunosuppressants. Although these medications are costly and produce unpleasant side effects, adherence is critical to decrease complications, reduce readmissions, and ultimately increase quality of life and survival.

Adherence is complex, but ultimately, the final common pathway to adherence is human behavior. In pediatrics, adherence is largely dependent on parents. As the primary caregivers, they are responsible for ensuring children receive the prescribed therapy correctly. In a high-risk HSCT population, caregivers are isolated with their child due to infection risk and must manage challenging treatment regimens at home, often with limited time and support. Complex behavioral interventions, typically employed to address adherence, are difficult to deliver and manage in the context of these daily tasks. Alternatively, behavioral economics (BE) theory suggests that small "nudges" can produce and sustain behavior change. A BE approach is a significant paradigm shift and assumes decision-making can be influenced through low-intensity interventions to lead patients to optimal choices. Improved adherence to medication and exercise programs using BE designed interventions in adults have been positive. Within pediatrics, BE has been successful in reducing childhood obesity, increasing vaccination rates, and improving adherence rates to infant HIV medications.

ELIGIBILITY:
Inclusion Criteria:

* Children of caregivers must be a) 0 to 21 years of age; b) receiving immunosuppression for an allogeneic transplant or anti-infective for an autologous transplant; c) discharged prior to Day 100 or completion of immunosuppression taper, and d) residing with the primary caregiver that enrolls on the study.
* Primary caregivers must be: d) English-speaking; and e) have an iOS or Android capable cellular device.

Exclusion Criteria:

* Adults unable to consent

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Momentary Event Monitoring System (MEMS) Caps | Baseline to day 100
  MEMS Caps collect daily data via a micro-electronic circuit that registers the opening and closing of the threaded pill bottle. Each opening and closing is assumed to reflect an administered and consumed medication dose. This data will be collected either at weekly or monthly from participants at their visits in the BMT clinic as a direct measure of adherence. Electronic monitors contain micro-electronic circuits that date and time-stamp each time the container is opened to remove a dose of medication. Data from the electronic monitors will be downloaded using cloud or computer-based software, at each study visit.53,54 An adherence percentage was calculated by dividing the number of doses taken by the number of doses prescribed for each day. All of the electronic monitors have been independently tested for accuracy.55
Medication Adherence Measure (MAM) | Baseline to day 100
  The MAM is semi-structured interview specific to pediatrics, conducted with the parent, to obtain an individual score in each module. The score is represented in percentages of the number of required doses. A total summary score can be calculated across all medications, as well as separately. This allows for quantification of the degree of adherence on a continuum. MAM has demonstrated adequate convergent validity with MEMs caps (r =-.40, p < .05).
System Usability Scale | Exit (Day 100)
  The SUS is a 10-item questionnaire routinely used to evaluate the functionality and acceptability of mHealth apps. Items are rated on a 5 point scale and scores range from 0 to 100. Reliability (0.91) and validity (.81 correlation with 7- point scale of "user friendliness") have been well established. A score of > 68% is considered above average.
Posttransplant Perception Survey | Baseline (Week 0)
  The posttransplant perception survey is a self-report clinical assessment tool adapted from the kidney transplant population for this trail. The tool contains 4 items asking participants to report on their views about their child's health and perceptions post-transplant. Items are rated on a 5 point Likert scale.
Barrier Assessment Tool | Baseline (Week 0)
  The Barrier Assessment Tool (BAT) is a self-report clinical assessment tool. The tool contains 14 commonly endorsed barriers with a checkbox next to each item. Domains include logistical issues (e.g., forgetting, inconvenience), ingestion difficulties (e.g., swallowing, taste), efficacy (e.g., feel I don't need it), financial difficulties, regimen characteristics (e.g., too many medications, side effects), and patient-specific issues (e.g., refusal by child, embarrassment). A sum total of the number of barriers is calculated, as well as concordance between caregiver and patient report. In the feasibility study, the average concordance between caregiver and patient report of each barrier (n=48) was 0.299.53 The total barrier score will be used. A sum total of 0 to 14 could be calculated, with higher scores indicating more barriers.
Caregiver Satisfaction | Exit (Day 100)
  Satisfaction will be assessed via semi-structured interviews and an electronic version of the Caregiver Satisfaction Questionnaire with caregivers. Caregivers will be asked for feedback regarding participation in the intervention, benefit, burden, barriers, suggested modifications, and overall satisfaction. Suggested modifications to the app and advice to the healthcare team will also be solicited. Due to the qualitative nature of the interview, caregiver responses cannot be scored but will be coded for themes. Questions on the Caregiver Satisfaction Questionnaire are scored on a 1 to 4 Likert scale with higher total scores indicating higher caregiver satisfaction.
Pediatric Quality of Life Inventory (PedsQL) version 4.0 | Week 3, Week 6, and Week 9
  Parents will complete the Pediatric Quality of Life Inventory (PedsQL) every three weeks (at week 3, week 6, and week 9). The frequency of 23 problems in 4 domains (i.e., physical, emotional, social, school) are rated on a 3 or 5-point scale. Versions are based on child age: (a) 5-7, (b) 8-12 and, (c) 13-18 years old.
Medy Remote Patient Management (RPM) medication box by Vaica | Baseline to day 100
  Medy RPM collects daily data via an NFC reader. Each opening and closing is assumed to reflect an administered and consumed medication dose. This data will be collected monthly from participants as a direct measure of adherence. Electronic monitors contain micro-electronic circuits that date and time-stamp each time the container is opened to remove a dose of medication. Data from the electronic monitors will be downloaded using cloud or computer-based software, at each study visit. An adherence percentage was calculated by dividing the number of doses taken by the number of doses prescribed for each day. All of the electronic monitors have been independently tested for accuracy.

SECONDARY OUTCOMES:
Demographic Data Form | Baseline (Week 0)
  The demographic data form is a questionnaire used to evaluate basic background characteristics including parent and child age, sex, race, ethnicity, education level, and family income.
Medication Possession Ratio (MPR) | Monthly until day 100
  MPR is a standard adherence measure that uses pharmacy refill records to calculate adherence using the sum of the days' supply obtained between the first pharmacy fill and the last fill divided by the total number of days. Higher scores indicate better adherence. The number of refills increases accuracy of the adherence estimate.
Medication Level Variability Index (MLVI) | Weekly until day 100
  The MLVI is the calculation of the standard deviation of serum assays of immunosuppressants that has shown to correlate with adherence and clinical outcomes in the solid organ transplant population.54 Immunosuppressant serum assays are collected weekly during the acute phase. A calculation of the degree of variation among levels will be formulated.
Graft vs. Host Disease (GVHD) | Weekly until day 100
  GVHD will be assessed on the international standard acute GVHD grading and staging scale. Provider grading will be per organ system on a 1-4 scale, with an overall score given weekly.
Readmissions | Weekly until day 100
  Readmission rates will be determined by the number of admissions requiring greater than a 24-hour stay within the first 100 days after discharge. Reason for readmission will be recorded and based on the EMR discharge diagnosis. In addition, a sub-analysis of readmissions within the first 30 days after initial discharge post-HSCT will be completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No